CLINICAL TRIAL: NCT03824015
Title: Keeping Adults Physically Active: Randomised Controlled Feasibility Study
Brief Title: Keeping Adults Physically Active Feasibility Study
Acronym: KAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16001; 16/LO/0396 (Other: London-Chelsea Health Research Authority)
Record Dates: First submitted 2019-01-14; First posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Physical Activity; Falls Prevention
Keywords: Physical Activity; Older Adults; Behaviour maintenance; feasibility study; falls prevention
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Six sessions of motivational interviewing over a six-month period. KAPA intervention sessions were held in accessible, community venues located within the local authorities of Derby City, Leicestershire and Rutland Counties. The KAPA intervention was delivered face-to-face by Postural Stability Instructors, in a group setting, using motivational interviewing. Sessions lasted between 60 to 90 minutes. Postural Stability Instructors delivered KAPA intervention sessions by telephone if a participant did not, or was unable to, attend a face-to-face session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KAPA intervention arm (Experimental): KAPA participants who completed the 24-week commissioned Falls Management Exercise program received six sessions of motivational interviewing over a six-month period. KAPA intervention sessions were held in accessible, community venues located within the local authorities of Derby City, Leicestershire and Rutland Counties. The KAPA intervention was delivered face-to-face by Postural Stability Instructors, in a group setting, using motivational interviewing. Sessions lasted between 60 to 90 minutes. Postural Stability Instructors delivered KAPA intervention sessions by telephone if a participant did not, or was unable to, attend a face-to-face session.
  Interventions: Behavioral: Keeping Adults Physically Active (KAPA) intervention
- Usual care (Other): The usual care participants finished the original Falls Management Exercise program and went on to being offered the service provider's usual care package.
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Keeping Adults Physically Active (KAPA) intervention — The Keeping Adults Physically Active (KAPA) intervention included six 60-90 minute group motivational interviewing sessions which were supported by a pedometer and a file containing information about locally run physical activity services, a home exercise booklet and written information on different types of lifestyle and transport related physical activity. During sessions the KAPA participants created physical activity plans and reflected on their physical activity diaries and personal physical activity goals. Various sub-sets of behaviour change techniques were delivered to help support the participants in continuing to be active.
  Arms: KAPA intervention arm
Other: Usual Care — Usual care was delivered for the duration of the KAPA feasibility study. The usual care participants finished the original Falls Management Exercise program and went on to being offered the service provider's usual care package. Upon initiating the KAPA feasibility study it was unknown what the service provider would deliver as usual care. Therefore a study objective was to describe the usual care package delivered by the service providers.
  Arms: Usual care

SUMMARY:
The Keeping Adults Physically Active (KAPA) feasibility study aimed to examine the feasibility and acceptability of the an intervention designed to encourage the continuation of physical activity following the completion of a Falls Management Exercise program.

DETAILED DESCRIPTION:
Background and premise:

Research shows that the continuation of physical activity wanes, and the positive health effects diminish, between eight-to-twelve months after the completion of community-based physical activity programs. A key finding of the Pro-Act 65 trial was that 24-months after the trial ended the beneficial effects of the Falls Management Exercise program diminished in the older people who reverted back to their old physical activity behaviours. Sustaining physical activity levels after the end of a structured physical activity program is critical to maintain any gains in functional status and falling risk. Furthermore, sustaining changes in physical activity behaviour is vital to the cost-effectiveness of physical activity interventions and to improve public health outcomes. Yet, little is known about what intervention components work best to promote the continuation of new physical activity behaviours once structured exercise programs have ceased. This suggests there is substantial opportunity to maintain the health and wellbeing of older people by implementing interventions that encourage the maintenance of physical activity.

The investigators have developed a complex evidence-based intervention that aims to engage older adults in positive physical activity behaviours after the completion of the Falls Management Exercise program. The intervention developed is based on the findings of a systematic review [PROSPERO registration: CDR42016038137] of physical activity maintenance interventions delivered to people aged 65 years and older and a review of national expert guidance on behaviour change. The intervention will be delivered to people who are exiting a 24-week community based Falls Management Exercise program within Leicestershire, Rutland Counties and Derby City and will be investigated in a feasibility trial.

The ProAct65+ trial shows that physical activity can be maintained for 12 months after the cessation of a Falls Management Exercise program. Data will be collected directly after the completion of the maintenance intervention which is also the six month time-point after the completion of the FaME program. Therefore it is possible that both the control and the intervention group may maintain their physical activity levels after the Falls Management Exercise program has ceased. Although maintenance may be higher in the intervention group, the treatment effect of the KAPA intervention will not be assessed due to the given timeframe of this study. However the feasibility trial will be used to collect the crucial data needed to inform a subsequent randomised control trial.

Study design:

The feasibility of the KAPA intervention was investigated in a two-arm, cluster randomised (clustering at the level of Postural Stability Instructor), multisite feasibility trial comparing the KAPA intervention with usual care controls conducted in 8 Falls Management Exercise classes nested within the PHysical activity Implementation Study In Community-dwelling AduLts (PHiSICAL) study.

Research Participants:

There were two types of study participants:

1. Community dwelling Falls Management Exercise program service users aged 65 years or older (referred to as KAPA participants).
2. Postural Stability Instructors who delivered Local Authority-commissioned Falls Management Exercise program in Derby City, Rutland or Leicestershire Counties (referred to as Postural Stability Instructors).

Intervention procedures:

KAPA participants who completed the 24-week commissioned Falls Management Exercise program received six sessions of PA motivational interviewing over a six-month period. KAPA intervention sessions were held in accessible, community venues located within the local authorities of Derby City, Leicestershire and Rutland Counties. The KAPA intervention was delivered face-to-face by Postural Stability Instructors, in a group setting, using motivational interviewing. Sessions lasted between 60 to 90 minutes. Postural Stability Instructor's delivered KAPA intervention sessions by telephone if a participant did not, or was unable to, attend a face-to-face session.

Control arm: Service providers usual care package.

The feasibility of the KAPA intervention was assessed by:

Objective 1: Feasibility of the research methods were assessed by estimating the recruitment and retention rates of the Postural Stability Instructors and the Falls Management Exercise program recipients to participate in the feasibility study.

Objective 2: Feasibility of the KAPA intervention was assessed by attendance rates and telephone response rates to the KAPA intervention as recorded in the class registers.

Objective 3: Assessing acceptability of the KAPA intervention by:

* Conducting semi-structure interviews with the participants in receipt of the intervention and the Postural Stability Instructors delivering the intervention, to assess the acceptability of the intervention features and delivery modes.
* To investigate the acceptability of the KAPA training day to the Postural Stability Instructors via a training evaluation questionnaire.

Objective 4: Investigating intervention adherence by:

* Analysing the Postural Stability Instructors completion rates of the class registers.
* Evaluating whether the participants completed the physical activity diaries and achieved their physical activity goals as recorded in the monthly class registers.
* The KAPA participants were also asked whether they adhered with the KAPA intervention during semi-structured interviews.

Objective 5: Assessing fidelity through:

* Observations of the initial consultations and group sessions.
* Postural Stability Instructors were asked whether they made any modifications to the KAPA intervention during a semi-structured interview.

Objective 6: Investigating parameter estimates of moderate to vigorous physical activity, the usual care descriptive and a data collection tool to cost the KAPA intervention for a future definitive trial by:

* Estimating the potential effect size of moderate to vigorous physical activity and percentage of the KAPA participants meeting the recommended 150 minutes of moderate to vigorous physical activity per week between the KAPA intervention and usual care arms.
* Estimating the intraclass correlation coefficient for moderate to vigorous physical activity using the Phone-FITT questionnaire.
* Usual care was described by its intervention features, delivery modes and the behaviour change strategies included.
* Identifying tools and testing the feasibility of collecting the data needed to cost the KAPA intervention to enable a cost-effective analysis in a definitive trial.

Objective 7: Recording adverse events and assessing them for causality to determine if they are related to the delivery of the KAPA intervention.

ELIGIBILITY:
Postural Stability Instructor participants

Inclusion criteria:

* Postural Stability Instructors in Leicestershire, Rutland or Derby City who were delivering a Local Authority-commissioned Falls Management Exercise program and were participating in the PHysical activity Implementation Study In Community-dwelling AduLts (PHiSICAL)study.
* Able to provide written informed consent.

Exclusion criteria:

* Postural Stability Instructors delivering a falls prevention programme or Falls Management Exercise program that was not commissioned within Derby City, Rutland or Leicestershire Counties and not participating in the PHysical activity Implementation Study In Community-dwelling AduLts (PHiSICAL) study.
* Unable to provide written informed consent

KAPA participants

Inclusion criteria:

* Enrolled on a Local Authority Falls Management Exercise program in Derby City, Rutland or Leicestershire Counties and participating in the PHysical activity Implementation Study In Community-dwelling AduLts (PHiSICAL) study.
* Able to provide written informed consent.

Exclusion criteria:

* Enrolled on a falls prevention programme or Falls Management Exercise program that was not commissioned within Derby City, Rutland or Leicestershire Counties and not participating in the PHysical activity Implementation Study In Community-dwelling AduLts (PHiSICAL) study.
* Unable to provide written informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-01-05 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention rates in the intervention and control group | 6 months
  The researchers recorded the number of study sites, Postural Stability Instructors and KAPA participants invited and recruited into the feasibility study. Retention rates were recorded as the number of KAPA participants (i.e. intervention and usual care participants) who remained within the study and provided outcome data at the 6-month time point.
Attendance rates to the KAPA intervention sessions | 6 months
  The Postural Stability Instructors documented in the class registers the KAPA participants' attendance at each of the monthly telephone or face-to-face community based KAPA intervention sessions. Class registers were used to record the number of face to face and telephone interactions with the participants.
Assessing acceptability of the KAPA intervention: semi-structure interviews | 12 months
  Acceptability of the intervention was determined via semi-structure interviews with the participants in receipt of the intervention and the Postural Stability Instructors delivering the intervention, to assess the acceptability of the intervention features and delivery modes. Interview data was analysed using a framework analysis approach.

SECONDARY OUTCOMES:
Training evaluation of the KAPA training day | 1 day
  After receiving KAPAs training the Postural Stability Instructors completed a training evaluation form to assess the suitability and acceptability of the training content and materials.
Adherence to key KAPA intervention strategies | 6 months
  The KAPA participant's adherence to the KAPA intervention was measured via completion of the physical activity diaries and achievement of monthly physical activity goals. The Postural Stability Instructors asked the participants if they had completed their diaries and achieved their goals during each face to face or telephone delivered KAPA intervention session. Participant responses were recorded by hand as a yes/no in the monthly class registers by the Postural Stability Instructors.
Fidelity of the KAPA interventions delivery | 6 months
  Fidelity was assess via observations of the KAPA sessions, which were recorded on a fidelity checklist.
Parameter estimates of moderate to vigorous physical activity and Intra Class Coefficient | 6 months
  Moderate to vigorous physical activity were collected using the Frequency Intensity Time Type (Phone-FITT) questionnaire at baseline and the 6-month time point.
  The Phone-FITT questionnaire measures household, recreational and seasonal activities. It does not provide a scoring system to categorise physical activity intensity as being light, moderate or vigorous. The Phone-FITT scoring system was re-categorised in terms of physical activity intensity across all household, recreational and seasonal physical activity in accordance with the Chief Medical Officers physical activity guidelines.
  The Phone-FITT questionnaire utilises ranges to estimate physical activity duration (e.g. 1-15 minutes). To calculate minutes of moderate to vigorous physical activity the median number within each range was coded to estimate minutes of weekly physical activity. Frequency was recorded in its absolute values (i.e. x3 week).
Defining usual care | 6 months
  A interview survey approach was used to collect the data relating to usual care. The aim was to describe usual care according to the following key elements:
  * Provide a brief description of usual care
  * Describe the type of PA behaviours did usual care targeted.
  * Describe the materials used to help deliver usual care.
  * Description of the usual care procedures and supporting activities.
  * Describe who delivered usual care.
  * Describe the modes of delivery.
  * Describe the location were the intervention was delivered.
  * Provide details on the duration, frequency, intensity and number of contacts that usual care was delivered.
  * Provide any details on tailoring or modifications to usual care. The researcher asked the Postural Stability Instructors open questions (either face to face or via phone) relating to each of these elements. The researcher completed the data collection form with the Postural Stability Instructors responses.
Developing a cost proforma to cost KAPA for a definitive trial | 9 months
  Data relating to how much it cost to deliver the KAPA intervention was collected using cost proformas completed by the service providers (i.e. Postural Stability Instructors and their managers). Cost proformas collected data on the costs incurred by the service providers to deliver the KAPA intervention. The data collected from the providers included costs relating to staff wages, travel expenses, administration costs, venue hire, consumables and expenses incurred to attend the training day. In addition a researcher recorded the research costs incurred to deliver the training day (i.e. venue hire, training manuals, trainer wages and trainer travel expenses).
The number of adverse events incurred in the KAPA intervention group. | 6 months
  All adverse events were recorded and monitored by the research team.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Orton, Principal Investigator — University of Nottingham and NIHR

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568
- [Derived] Audsley S, Kendrick D, Logan P, Jones M, Orton E. A randomised feasibility study assessing an intervention to keep adults physically active after falls management exercise programmes end. Pilot Feasibility Stud. 2020 Mar 7;6:37. doi: 10.1186/s40814-020-00570-9. eCollection 2020. PMID 32161660